CLINICAL TRIAL: NCT06616077
Title: Determinaton of Changes in the Endometrial Gene Expression Profile Induced by Exogenous Progesterone After Post-ovulatory Administration of Mifepristone
Brief Title: Endometrial Transcript Profile with Progesterone After Post-ovulatory Mifepristone
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Reproductive Health Research Insritute, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RU001
Record Dates: First submitted 2024-09-17; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Endometrial Endocrine Regulation; Progesterone Supplementation in Women After Mifepristone
Keywords: Endometrial gene expression; Progesterone; Mifepristone; RU486; Secretory endometrium
MeSH Terms: interventions — Progesterone; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mife + PLA (Placebo Comparator): Oral mifepristone 200 mg two days after positive LH (LH+2) and vaginal placebo during LH+3 until LH+5
  Interventions: Drug: mifepristone 200 mg; Drug: Placebo Vaginal
- Mife + P4 (Experimental): Oral mifepristone 200 mg two days after positive LH (LH+2) and vaginal micronized progesterone (600 mg/day) during LH+3 until LH+5
  Interventions: Drug: Micronized Progesterone 600 mg; Drug: mifepristone 200 mg
- PLA + P4 (Active Comparator): An oral placebo pill two days after positive LH (LH+2) and vaginal micronized progesterone (600 mg/day) during LH+3 until LH+5
  Interventions: Drug: Micronized Progesterone 600 mg; Drug: Oral Placebo Tablet
- PLA + PLA (Placebo Comparator): An oral placebo pill two days after positive LH (LH+2) and a vaginal placebo during LH+3 until LH+5
  Interventions: Drug: Oral Placebo Tablet; Drug: Placebo Vaginal

INTERVENTIONS:
Drug: Micronized Progesterone 600 mg — Vaginal supplementary micronized progesterone will be given after postovulatory administration of the progesterone receptor antagonist mifepristone. Administration from LH+3 to LH+5 (LH peak=LH+0); 200 mg 3 times per day.
  Other Names: Progendo
  Arms: Mife + P4; PLA + P4
Drug: mifepristone 200 mg — Post ovulatory single oral administration (LH+2, LH peak=LH+0)
  Other Names: MIFEAPROFA
  Arms: Mife + P4; Mife + PLA
Drug: Oral Placebo Tablet — Oral placebo tablet containing brewer yeast, cellulose, stearic acid, silica, magnesium stearate
  Arms: PLA + P4; PLA + PLA
Drug: Placebo Vaginal — Cocoa butter
  Arms: Mife + PLA; PLA + PLA

SUMMARY:
The goal of this exploratory trial is to determine the endometrial gene expression profile induced by exogenous progesterone after postovulatory administration of mifepristone. It will also learn about the plasticity ofr the endometrial response to progesterone. The main questions it aims to answer are:

Is exogenous progesterone able to modulate the gene expression of endometrial transcripts that have been altered by mifepristone?

Researchers will compare the endometrial gene expression profiles with exogeonous progesterone to a placebo (a look-alike substance that contains no drug) after postovulatory administration of mifepristone.

Participants will:

Do ovulation follow-up tests at home assesing LH in urine Visit the hospital 2 days after a positive LH for mifepristone administration and ultrasonography check of ovaries and uterus.

Starting from the next day, take progesterone or placebo for 3 days. Visit the hospital 2 days after that for ultrasonography check of ovaries and uterus and for an endometrial and blood sample collection.

The endometrial samples will be processed to isolate the RNA and for histological assessment. Gene expression profiles will be determined by RNA-seq.

DETAILED DESCRIPTION:
Objective: To determine the effect of progesterone supplementation on the mid-secretory endometrial transcript profile after postovulatory administration of mifepristone.

Design: A randomized, double-blind, placebo-controlled study. Setting: Tertiary academic medical center Subjects: A total of 9 Hispanic women of proven fertility who had been surgically sterilized.

Interventions: Participating women received a single dose of mifepristone 200mg 48 hours after the LH peak (LH+2, LH+0=LH peak). Endometrial samples were obtained on LH+7 after vaginal administration of micronized progesterone (600mg/day) for 3 days (LH+3 to LH+5). Each woman contributed with one cycle treated with placebo and another with progesterone (group A). Additionally, endometrial samples were obtained on LH+7 from subset of 4 women who did not receive mifepristone; with each one contributing with one cycle treated with vaginal progesterone supplementation or placebo as a reference (group B). Endometrial thickness, circulating progesterone levels, and endometrial histology were also documented in all cycles. RNA-seq was used to identify genes whose transcript levels significantly changed by the administration of progesterone versus placebo, with postovulatory administration of mifepristone. The transcript profiles of these genes were further evaluated in the endometrial samples from group B.

ELIGIBILITY:
Inclusion Criteria:

* proven fertility
* regular menstrual cycles
* surgically sterilized at least one year before participating in the protocol

Exclusion Criteria:

* chronic medical problems
* abnormal results of screening blood tests
* ovarian masses
* symptomatic endometriosis
* uterine leiomyomata
* being under chronic medication or taking hormones or drugs able to modify the metabolism of steroid hormones in the 3 preceding months to study enrollment

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Endometrial Gene Expression Profile | From enrollment to the end of treatments after aproximately 12 weeks
  RNA-seq gene expression in the midluteal phase

SECONDARY OUTCOMES:
Endometrial dating | From enrollment to the end of treatments after aproximately 8 months
  Estimated cycle day based on endometrial morphology according to the Noyes criteria

OTHER OUTCOMES:
Uterine ultrasonographic features | From enrrollment to the end of treatments after 12 weeks
  Will be evaluated the ultrasonographic features such as hypo- and hyper- echogenecity
Circulating progesterone levels | From enrollment to after the treatments after 12 weeks
  Will be evaluated the cirduating levels of progesterone on day LH+7 (LH+0=LH peak) in women that have taken postovulatory mifepristone plus exogenous progesterone or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro A Tapia-Pizarro, Biologist, PhD, Study Director — University of Chile
Locations (1):
- Hospital San Borja Arriarán, Santiago, Santiago Metropolitan, Chile